CLINICAL TRIAL: NCT04782843
Title: Evaluation of the Intra-observer Agreement of the HEP Score in Surgical Intensive Care.
Acronym: REPROHEP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/586
Record Dates: First submitted 2021-03-02; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Heparin-induced Thrombocytopenia
Keywords: Heparin-induced Thrombocytopenia; HEP score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: he retrospective cohort studied includes all the patients included in a previous study carried out in our center, the objective of which was to study the diagnostic performance of the HEP score in surgical intensive care.
  The cohort studied is made up of all patients admitted for surgical resuscitation between October 2011 and October 2013 and validating the following criteria:
  * Inclusion criteria: any adult patient (age ≥ 18 years), admitted to surgical intensive care, treated with heparin (UFH or LMWH), and suspected of TIH by a clinician in the department according to the criteria of the SFAR 2002.
  * Non-inclusion criteria: minor patients, pregnant women and adults incapable.
  Interventions: Other: HEP score assessement

INTERVENTIONS:
Other: HEP score assessement — Assessement of the HEP score between 2 physician.

SUMMARY:
The main objective of this work is to assess the intraoperator reproducibility in the calculation of the HEP score in a population of intensive care patients.

DETAILED DESCRIPTION:
The "HEP score" (HIT Expert Probability) is also a clinical probability score, created thanks to the experience of clinicians (16). It is very recent and therefore still little studied and little used. In particular, it has not been the subject of a prospective validation study for ICU patients.

The use of this score is therefore not recommended in everyday practice.

However, the literature shows a higher diagnostic value of the HEP score especially for resuscitation-type patients, as well as when used by an operator with little experience. This could be due to greater detail given in consideration of other causes of thrombocytopenia (17).

The main objective of this work is to assess the intraoperator reproducibility in the calculation of the HEP score in a population of intensive care patients.

The secondary objectives will aim to:

* Evaluate inter-operator reproducibility
* Determine if the reproducibility of the HEP score is influenced by:

The patient's sex The type of heparin used (LMWH vs UFH) The severity of the patient (IGS2 score) A history of cardiac or orthopedic surgery

The expected consistent benefits allow validation of the HEP score in surgical intensive care (cf. EVHEP-TIH study).

This would allow a better assessment of the pre-test probabilities of TIH with the performance of biological tests.

ELIGIBILITY:
Inclusion Criteria:

* any adult patient (age ≥ 18 years), admitted to surgical intensive care, treated with heparin (UFH or LMWH), and suspected of TIH by a clinician in the department according to the criteria of the SFAR 2002.

Exclusion Criteria:

* Non-inclusion criteria: minor patients, pregnant women and adults incapable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort studied is made up of all patients admitted for surgical resuscitation between October 2011 and October 2013
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Intraobserver agreeement for the HEP score | 3 months
  Intraobserver agreeement for the HEP score

SECONDARY OUTCOMES:
Interobserver agreement for the HEP score | 3 months
  Interobserver agreement for the HEP score

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Besch, MD, Principal Investigator — CHRU J. Minjoz à Besançon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cuker A, Arepally G, Crowther MA, Rice L, Datko F, Hook K, Propert KJ, Kuter DJ, Ortel TL, Konkle BA, Cines DB. The HIT Expert Probability (HEP) Score: a novel pre-test probability model for heparin-induced thrombocytopenia based on broad expert opinion. J Thromb Haemost. 2010 Dec;8(12):2642-50. doi: 10.1111/j.1538-7836.2010.04059.x. PMID 20854372
- See also: Princeps article — https://pubmed.ncbi.nlm.nih.gov/20854372/